CLINICAL TRIAL: NCT00492011
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Ability of Ramelteon 1 mg, 4 mg, and 8 mg to Alleviate the Insomnia Symptoms Associated With Eastward Bound Jet Lag Across 5 Time Zones in Healthy Adult Volunteers
Brief Title: Efficacy of Ramelteon on Insomnia Symptoms Associated With Jet Lag in Healthy Adult Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-375-045; U1111-1115-1566 (Registry Identifier: WHO)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Circadian Dysregulation
Keywords: Circadian Rhythm Disorders; Biological Clock Disturbances; Jet Lag Syndrome; Time Zone Change Syndrome; Drug Therapy
MeSH Terms: conditions — Chronobiology Disorders; Jet Lag Syndrome | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ramelteon 1 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 4 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 1 mg, tablets, orally, once nightly for 4 nights.
  Other Names: TAK-375; Rozerem™
  Arms: Ramelteon 1 mg QD
Drug: Ramelteon — Ramelteon 4 mg, tablets, orally, once nightly for 4 nights.
  Other Names: TAK-375; Rozerem™
  Arms: Ramelteon 4 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once nightly for 4 nights.
  Other Names: TAK-375; Rozerem™
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once nightly for 4 nights.
  Arms: Placebo

SUMMARY:
The purpose of this study to determine the degree to which ramelteon, once daily (QD), can reduce the insomnia symptoms associated with rapid, eastward travel across 5 time zones.

DETAILED DESCRIPTION:
Circadian dysrhythmia, or jet lag, is defined as multiple biologic and psychologic stresses created by rapid travel across multiple time zones. As more people are transported by jet aircraft, the issue of jet lag becomes more important. What was an inconvenience during travel for leisure is now a physiologic consequence for the travelers and crew.

Jet lag is composed of a variety of unpleasant symptoms that vary with the number of time zones crossed, the individual, and even the direction flown (east versus west). The most typical symptoms include daytime sleepiness, fatigue, impaired alertness, and trouble initiating and maintaining sleep. Other symptoms of circadian dysrhythmia are insomnia, gastrointestinal complaints, apathy, weakness, irritability, malaise, and loss of appetite. Travel across time zones also has been associated with diabetic ketoacidosis, depression, and impaired cognitive performance in individuals at risk. Decreased sport performance has been noted in several studies.

In addition to environmental and social cues, physical factors, such as age, hydration status, and illness, could adversely affect the ability to entrain (adjust) quickly. The stressors of flight, noise, vibration, decreased humidity, barometric pressure changes, and decreased partial pressure of oxygen all contribute to crew and travelers health at the destination.

Being out of synchronicity with the environment causes jet lag symptoms. Travel through time zones places the body in a situation when it must sleep when not tired and awaken when the internal cues are initiating sleep. The brain's internal clock is the suprachiasmatic nucleus within the hypothalamus the body is in a constant state of circadian adjustment to remain entrained to a given time zone. In addition to the subjective feeling of well being are measurable changes associated with daily patterns. For example, core body temperature changes throughout the day and decreases before falling asleep. Melatonin levels increase in the evening and night and recede during the day.

Ramelteon is a melatonin receptor 1 and melatonin receptor 2 agonist currently marketed in the US for the treatment of insomnia characterized by difficulty with sleep onset. Study participation is anticipated to be about 2 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Willing to travel from Hawaii to the East Coast and have a minimum stay of 6 days at the destination in a sleep laboratory during the entire study.
* Has lived in Hawaii for at least 12 months and has not been traveling outside of Hawaii for 4 consecutive days within 30 days prior to the Outpatient Screening Visit.
* History of sleep disturbance associated with jet lag symptoms, with at least two occurrences in the last three years, as defined in the International Classification of Sleep Disorders.
* Habitual bedtime should be determined by sleep history as between 9:00 PM and 12:00 AM as determined by sleep history prior to randomization.
* Have regular bedtime (within 1 hour) for 1 week prior to travel.
* The subject has a subjective sleep latency of less than 30 minutes and a subjective total sleep time of 6.5 hours but less than 9 hours, as determined by sleep history.
* Mean subjective sleep latency of less than 30 minutes and a mean subjective total sleep time of greater than 6.5 hours but less than 9 hours in 3 of 5 nights after the outpatient screening visit, as determined by post-sleep questionnaire.
* Willingness and ability to comply with study procedures, including travel time, sleep, and waking-hour activities, light-exposure restriction, and food intake.
* Body mass index between 18 and 34, inclusive.
* Negative test result for selected substances of abuse (including alcohol) at Initial Screening, the In-Patient Actigraphy Screening Nights 1 and 2, and the Treatment Period.
* Negative test result for hepatitis B Surface antigen and hepatitis C virus antibody.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin, and melatonin related compounds.
* History of primary sleep disorders as determined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised within the past 6 months.
* Current sleep disorder as assessed by presence of sleep apnea, period leg movement syndrome, insomnia, daytime napping of more than 20 minutes, chronic fatigue.
* Ever had a history of seizures, sleep apnea, restless leg syndrome, periodic limb movement syndrome, or chronic obstructive pulmonary disease.
* History of psychiatric disorder (including schizophrenia, bipolar disorder, mental retardation, or cognitive disorder, anxiety, or depression) within the past 12 months.
* Current, clinically significant neurological (including cognitive), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, or metabolic disease, as determined by the investigator.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised, or regularly consumes more than 14 alcoholic drinks per week.
* History of drug abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised.
* Positive urine drug screen or a positive urine drug screen or alcohol breathalyzer test.
* Sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the administration of single blind study medication.
* Positive hepatitis panel including anti- hepatitis A virus (only IgM is exclusionary), hepatitis B surface antigen, or anti- hepatitis C virus.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * cause a situation such that it would not be in the best interest of the subject to participate in the study.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the administration of study medication.
* Smokes greater than 3 cigarettes per day or uses tobacco products during nightly awakenings.
* Has flown across greater than 3 time zones within 28 days prior to or during screening.
* Reports high caffeine consumption (greater than 600 mg daily).
* Participated in any other investigational study and/or taken any investigational drug within 30 days or 5 half-lives of the investigational drug prior to the first dose of double blind study medication, whichever is longer.
* Used any central nervous system medication within 1 week (or 5 half lives of the drug, whichever is longer) prior to the administration of study medication. These medications must not have been used to treat psychiatric disorders.
* Used prescription or over-the-counter (OTC) hypnotic medication (including melatonin) within 3 months of the screening visits.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Anxiolytics
  * Sedatives
  * Antidepressants
  * CNS active drugs (including herbal)
  * Anticonvulsants
  * Narcotic analgesics
  * Sedating H1 antihistamines
  * St. John's Wort
  * Systemic steroids
  * Kava-kava
  * Respiratory stimulants
  * Ginkgo-biloba
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Antipsychotics
  * Over-the-counter and prescription diet aids
  * Muscle Relaxants Drugs affecting sleep/wake function
  * Melatonin
  * Modafinil

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2007-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Average Latency to Persistent Sleep measured by polysomnography. | Nights 2, 3, and 4

SECONDARY OUTCOMES:
Dim light melatonin offset time in a subset of subjects defined as the time of the morning when the melatonin drops to below 3 pg/mL with a downward slope. | Nights 2, 3, and 4
Total sleep time in minutes by polysomnography. | Nights 2, 3, and 4
Number of awakenings after persistent sleep by polysomnography. | Nights 2, 3, and 4
Wake time after persistent sleep onset by polysomnography. | Nights 2, 3, and 4
Sleep efficiency by polysomnography. | Nights 2, 3, and 4
Karolinska Sleepiness Scale | Days 1, 2, 3, 4 and 5
Pittsburgh Sleep Quality Index | Day 6
Daytime Function measured by Daytime Function Questionnaire (DTFQ) and Psychomotor Vigilance test (PVT) | Day 3
Digit Symbol Substitution Test | Days 1, 2, 3, 4 and 5
Memory Recall Test | Days 1, 2, 3, 4 and 5
Visual Analogue Scale for Mood and Feelings, level of alertness and ability to concentrate | Days 1, 2, 3, 4 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (4):
- United States (4):
  - Miami, Florida
  - Pembroke Pines, Florida
  - Honolulu, Hawaii
  - New York, New York

REFERENCES:
- [Result] Zee PC, Wang-Weigand S, Wright KP Jr, Peng X, Roth T. Effects of ramelteon on insomnia symptoms induced by rapid, eastward travel. Sleep Med. 2010 Jun;11(6):525-33. doi: 10.1016/j.sleep.2010.03.010. Epub 2010 May 18. PMID 20483660
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI